CLINICAL TRIAL: NCT01247285
Title: A Relative Bioavailability Study of 90 mg Fluoxetine Hydrochloride Capsules Under Non-Fasting Conditions
Brief Title: 90 mg Fluoxetine Hydrochloride Capsules Under Non-Fasting Conditions
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Teva Pharmaceuticals USA (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: R01-141
Record Dates: First submitted 2010-11-22; First posted 2010-11-24 (Estimated); Results first posted 2011-02-21 (Estimated); Last update posted 2011-02-21 (Estimated); Status verified 2011-01

CONDITIONS: Healthy
Keywords: Bioequivalence; Healthy Subjects
MeSH Terms: interventions — Fluoxetine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Investigational Test Product (Experimental): 90 mg Fluoxetine Hydrochloride Capsules (Teva)
  Interventions: Drug: Fluoxetine Hydrochloride
- Reference Listed Drug (Active Comparator): 90 mg PROZAC WEEKLY® Capsules (Eli Lilly)
  Interventions: Drug: PROZAC WEEKLY®

INTERVENTIONS:
Drug: Fluoxetine Hydrochloride — 90 mg Capsules
  Arms: Investigational Test Product
Drug: PROZAC WEEKLY® — 90 mg Capsules
  Other Names: Fluoxetine Hydrochloride (generic name)
  Arms: Reference Listed Drug

SUMMARY:
This study compared the relative bioavailability (rate and extent of absorption) of 90 mg Fluoxetine Hydrochloride Capsules by Teva Pharmaceuticals, USA with that of 90 mg PROZAC WEEKLY® Capsules by Eli Lilly and Company following a single oral dose (1 x 90 mg) in healthy adult volunteers under non-fasting conditions.

ELIGIBILITY:
Inclusion Criteria:

* Screening Demographics: All volunteers selected for this study will be healthy men or women 18 years or age or older at the time of dosing. The weight range will not exceed + 15% for height and body frame as per Desirable Weights for Men - 1983 Metropolitan Height and Weight Table or as per Desirable Weights for Women - 1983 Metropolitan Height and Weight Table.
* Screening Procedures: Each volunteer will complete the screening process within 28 days prior to Period I dosing. Consent documents for both the screening evaluation and HIV antibody determination will be reviewed, discussed, and signed by each potential participant before full implementation of screening procedures.
* If female and:

  * Of childbearing potential, is practicing an acceptable method of birth control for the duration of the study as judged by the investigator(s), or
  * Is postmenopausal for at least 1 year, or
  * Is surgically sterile (bilateral tubal ligation, bilateral oophorectomy, or hysterectomy).

Exclusion Criteria:

* Volunteers with a recent history of drug or alcohol addiction or abuse.
* Volunteers with the presence of a clinically significant disorder involving the cardiovascular, respiratory, renal, gastrointestinal, immunologic, hematologic, endocrine, or neurological system(s) or psychiatric disease (as determined by the clinical investigators).
* Volunteers whose clinical laboratory test values are outside the acceptable reference range and when confirmed on re-examination are deemed to be clinically significant.
* Volunteers demonstrating a positive hepatitis B surface antigen screen or a reactive HIV antibody screen.
* Volunteers demonstrating a positive drug abuse screen when screened for this study.
* Female volunteers demonstrating a positive pregnancy screen.
* Female volunteers who are currently breastfeeding.
* Volunteers with a history of allergic response(s) to fluoxetine or related drugs.
* Volunteers with a history of clinically significant allergies including drug allergies.
* Volunteers with a clinically significant illness during the 4 weeks prior to Period I dosing (as determined by the clinical investigators).
* Volunteers who currently use tobacco products.
* Volunteers who have taken any drug known to induce or inhibit hepatic drug metabolism in the 30 days prior to Period I dosing.
* Volunteers who report donating greater than 150 mL of blood within 30 days prior to Period I dosing. All subjects will be advised not to donate blood for 4 weeks after completing the study.
* Volunteers who have donated plasma within 14 days prior to Period I dosing. All subjects will be advised not to donate plasma for 4 weeks after completing the study.
* Volunteers who report receiving any investigational drug within 30 days prior to Period I dosing.
* Volunteers who report taking any systemic prescription medications in the 14 days prior to Period I dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2001-05; Primary Completion 2001-07 (Actual); Study Completion 2001-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: James D Carlson, Pharm.D., Principal Investigator — PRACS Institute, Ltd.
Locations (1):
- PRACS Institute, Ltd., Fargo, North Dakota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Fluoxetine Hydrochloride (Test) First: 90 mg Fluoxetine Hydrochloride Capsules test product dosed in first period followed by 90 mg Prozac® Weekly Capsules reference product dosed in the second period.
- Prozac® Weekly (Reference) First: 90 mg Prozac® Weekly Capsules reference product dosed in first period followed by 90 mg Fluoxetine Hydrochloride Capsules test product dosed in the second period.
Period: First Intervention
Arm/Group | Fluoxetine Hydrochloride (Test) First | Prozac® Weekly (Reference) First
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Washout of 28 Days
Arm/Group | Fluoxetine Hydrochloride (Test) First | Prozac® Weekly (Reference) First
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0
Period: Second Intervention
Arm/Group | Fluoxetine Hydrochloride (Test) First | Prozac® Weekly (Reference) First
Started | 13 | 13
Completed | 13 | 13
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Fluoxetine Hydrochloride (Test) First | Prozac® Weekly (Reference) First | Total
Number analyzed (Participants) | 13 | 13 | 26
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 13 | 13 | 26
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 4 | 10
  Male | 7 | 9 | 16
Race/Ethnicity, Customized [Number; unit: participants]
  Caucasian | 13 | 13 | 26
Region of Enrollment [Number; unit: participants]
  United States | 13 | 13 | 26

OUTCOME MEASURES:

1. Primary Outcome: Cmax of Fluoxetine.
Description: Bioequivalence based on Fluoxetine Cmax (maximum observed concentration of drug substance in plasma).
Time Frame: Blood samples collected over a 25 day period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Groups:
- Fluoxetine Hydrochloride (Test): 90 mg Fluoxetine Hydrochloride Capsules test product dosed in either period.
- Prozac® Weekly (Reference): 90 mg Prozac® Weekly Capsules reference product dosed in first either period.
Arm/Group | Fluoxetine Hydrochloride (Test) | Prozac® Weekly (Reference)
Number analyzed (Participants) | 26 | 26
ng/mL | 75.32 (14.7) | 69.86 (14.9)
Statistical Analysis 1: Comparison: Fluoxetine Hydrochloride (Test) vs Prozac® Weekly (Reference); Test type: Non-Inferiority or Equivalence — ANOVA is to be used to identify the source contributions by factors including subjects, period, formulation and potential interactions. The geometric mean ratio together with the ANOVA residual mean error term are used to identify the statistical basis for the 90% confidence interval for the ratio of the population means (Test [T]/Reference[R]) of the identified metrics (e.g. AUC, Cmax); Ratio of the T/R geometric mean x 100 = 107.81, 90% CI 2-sided [97.37 to 119.38] — Bioequivalence is established if the 90% confidence interval for the ln-transformed geometric mean between the reference (R) and test (T) product fall within the interval of 80-125%

2. Primary Outcome: AUC0-t of Fluoxetine.
Description: Bioequivalence based on Fluoxetine AUC0-t (area under the concentration-time curve from time zero to time of last measurable concentration).
Time Frame: Blood samples collected over a 25 day period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Fluoxetine Hydrochloride (Test) | Prozac® Weekly (Reference)
Number analyzed (Participants) | 26 | 26
ng*h/mL | 4148.71 (719.0) | 4120.11 (614.1)
Statistical Analysis 1: Comparison: Fluoxetine Hydrochloride (Test) vs Prozac® Weekly (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.69, 90% CI 2-sided [92.90 to 109.14] — [estimate comment as in outcome 1, analysis 1]

3. Primary Outcome: AUC0-inf of Fluoxetine.
Description: Bioequivalence based on Fluoxetine AUC0-inf (area under the concentration-time curve from time zero to infinity).
Time Frame: Blood samples collected over a 25 day period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Fluoxetine Hydrochloride (Test) | Prozac® Weekly (Reference)
Number analyzed (Participants) | 26 | 26
ng*h/mL | 4432.21 (1591.0) | 4398.46 (1277.0)
Statistical Analysis 1: Comparison: Fluoxetine Hydrochloride (Test) vs Prozac® Weekly (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 100.77, 90% CI 2-sided [93.53 to 108.56] — [estimate comment as in outcome 1, analysis 1]

4. Secondary Outcome: Cmax of Norfluoxetine.
Description: Informational comparison of Cmax values for the metabolite Norfluoxetine.
Time Frame: Blood samples collected over a 25 day period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Fluoxetine Hydrochloride (Test) | Prozac® Weekly (Reference)
Number analyzed (Participants) | 26 | 26
ng/mL | 35.11 (12.6) | 33.47 (13.1)
Statistical Analysis 1: Comparison: Fluoxetine Hydrochloride (Test) vs Prozac® Weekly (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 104.88, 90% CI 2-sided [98.53 to 111.64] — This analysis was for informational purposes only and was not used to establish bioequivalence

5. Secondary Outcome: AUC0-t of Norfluoxetine.
Description: Informational comparison of AUC0-t values for the metabolite Norfluoxetine.
Time Frame: Blood samples collected over a 25 day period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Fluoxetine Hydrochloride (Test) | Prozac® Weekly (Reference)
Number analyzed (Participants) | 26 | 26
ng*h/mL | 114575.21 (3451) | 10849.08 (2978)
Statistical Analysis 1: Comparison: Fluoxetine Hydrochloride (Test) vs Prozac® Weekly (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 105.64, 90% CI 2-sided [99.97 to 111.56] — This analysis was for informational purposes only and was not used to establish bioequivalence

6. Secondary Outcome: AUC0-inf of Norfluoxetine.
Description: Informational comparison of AUC0-inf values for the metabolite Norfluoxetine.
Time Frame: Blood samples collected over a 25 day period.
Population: All participants that completed the study had their samples analyzed.
Measure: Mean (Standard Deviation); unit: ng*h/mL
Arm/Group | Fluoxetine Hydrochloride (Test) | Prozac® Weekly (Reference)
Number analyzed (Participants) | 26 | 26
ng*h/mL | 13505.84 (5234) | 13365.13 (6325)
Statistical Analysis 1: Comparison: Fluoxetine Hydrochloride (Test) vs Prozac® Weekly (Reference); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 1]; Ratio of the T/R geometric mean x 100 = 101.05, 90% CI 2-sided [94.76 to 107.77] — This analysis was for informational purposes only and was not used to establish bioequivalence

ADVERSE EVENTS:
Time Frame: Adverse event data was collected over the course of the study, which was approximately 6 weeks in duration.
Description: Volunteers were monitored throughout the study for any adverse experiences. AEs were collected through both solicited and unsolicited methods. The volunteers were encouraged to report signs, symptoms, and any changes in health to the clinic staff.
Groups:
- Prozac® Weekly (Reference): 90 mg Prozac® Weekly Capsules reference product dosed in either period.
Arm/Group | Fluoxetine Hydrochloride (Test) | Prozac® Weekly (Reference)
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/26
Other Adverse Events (participants affected / at risk) | 11/26 | 11/26
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fluoxetine Hydrochloride (Test) (N=26) | Prozac® Weekly (Reference) (N=26)
Headache (General disorders) | 6 (8) | 6 (8)
Malaise (General disorders) | 2 (2) | 1 (1)
Nausea (General disorders) | 3 (4) | 2 (2)
Pharyngitis (General disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The Principal Investigator is not permitted to discuss or publish trial results.